CLINICAL TRIAL: NCT02203149
Title: A Phase II, Randomized Clinical Trial to Study the Safety, Tolerability, and Efficacy of the Combination Regimen of MK-5172 and MK-8742 in Japanese Subjects With Chronic Hepatitis C and a Phase III, Randomized Placebo-Controlled Clinical Trial to Study the Safety, Tolerability, and Efficacy of the Combination Regimen of MK-5172 and MK-8742 in Japanese Subjects With Chronic Hepatitis C
Brief Title: Study of Grazoprevir (MK-5172) and Elbasvir (MK-8742) in Japanese Participants With Chronic Hepatitis C (MK-5172-058)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5172-058; 142638 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2014-07-25; First posted 2014-07-29 (Estimated); Results first posted 2016-10-11 (Estimated); Last update posted 2018-09-24 (Actual); Status verified 2018-08

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Part 1 Grazoprevir 50 mg + Elbasvir (Experimental): Non-cirrhotic participants take 50 mg grazoprevir in combination with 50 mg elbasvir by mouth (p.o.) once daily (q.d.) for 12 weeks during the blinded period of Part 1 and are followed-up for 24 weeks during the open-label period of Part 1.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Placebo to Grazoprevir
- Part 1 Grazoprevir 100 mg + Elbasvir (Experimental): Non-cirrhotic participants take 100 mg grazoprevir in combination with 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 1 and are followed-up for 24 weeks during the open-label period of Part 1.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir (Experimental): Non-cirrhotic participants take grazoprevir (50 mg or 100 mg dose selected from Part I) and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2 and are followed-up for 24 weeks during the open-label period of Part 2.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir
- Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir (Placebo Comparator): Non-cirrhotic participants take dose-matched placebo p.o. q.d. for 12 weeks during the blinded period of Part 2 followed by a 4-week follow-up. Afterwards, participants take grazoprevir (50 mg or 100 mg dose selected from Part I) and 50 mg elbasvir p.o. q.d. for 12 weeks and are followed-up for 24 weeks during the open-label period of Part 2.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir; Drug: Placebo to Grazoprevir; Drug: Placebo to Elbasvir
- Part 2 Cirrhotic: Grazoprevir + Elbasvir (Experimental): Cirrhotic participants take grazoprevir (50 mg or 100 mg dose selected from Part 1) and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2, and are followed-up for 24 weeks during the open-label period of Part 2.
  Interventions: Drug: Grazoprevir; Drug: Elbasvir

INTERVENTIONS:
Drug: Grazoprevir — One or two 50 mg tablets (depending on randomization) taken orally once daily for 12 weeks.
Drug: Elbasvir — One 50 mg tablet taken orally once daily for 12 weeks.
Drug: Placebo to Grazoprevir — One tablet of placebo matched to grazoprevir, taken orally once daily for 12 weeks.
  Arms: Part 1 Grazoprevir 50 mg + Elbasvir; Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir
Drug: Placebo to Elbasvir — One tablet of placebo matched to elbasvir, taken orally once daily for 12 weeks.
  Arms: Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir

SUMMARY:
This is a two-part study of grazoprevir (MK-5172) + elbasvir (MK-8742) in Japanese participants with chronic hepatitis C virus (HCV) genotype 1 (GT1). Part I is a dose-finding study; in Part II, participants will be randomly assigned to receive grazoprevir at the dose determined in Part I in combination with elbasvir. The primary study hypothesis is that the percentage of treatment-naïve participants in the Immediate Treatment Arm of Part II who achieve sustained viral response at 12 weeks after the end of all treatment (SVR12) will be greater than the reference rate of 75%. A separate study arm for cirrhotic participants will also be included in Part II; these participants will receive grazoprevir at the determined dose in combination with elbasvir.

DETAILED DESCRIPTION:
In Part 1, HCV GT1 participants are randomized into one of two arms: 50 mg grazoprevir plus 50 mg elbasvir for 12 weeks during the double blinded (DB) period followed by 24 weeks of follow-up (FU) during an open-label (OL) period [Arm 1]; or 100 mg grazoprevir plus 50 mg elbasvir for 12 weeks during the DB followed by 24 weeks of FU during the OL [Arm 2]. Unblinding will occur after all participants complete FU Week 4 at which time the grazoprevir dose will be selected.

In Part 2, non-cirrhotic HCV GT1 participants and GT1 participants with compensated liver cirrhosis all receive the selected dose of grazoprevir (50 mg or 100 mg from Part 1) with 50 mg elbasvir for 12 weeks. Non-cirrhotic GT1 participants are randomized to receive either a) 12 weeks of active treatment immediately during the DB with 24 weeks of FU in the OL [Arm 1/Immediate Arm] or b) placebo for 12 weeks with 4 weeks of follow-up during the DB followed by 12 weeks of active treatment and 24 weeks of follow-up during the OL [Arm 2/Deferred Arm]. All cirrhotic participants [Arm 3/Cirrhotic] receive the selected dose immediately for 12 weeks during the DB with 24 weeks of FU during the OL.

Safety analyses for Part 1 and Part 2 arms will focus on the 12 week treatment phase plus the first 4 FU weeks. For the Part 2 Deferred Arm this will include the initial 12 week placebo treatment and first 4 weeks of FU. Efficacy analyses for Parts 1 and 2 will evaluate active treatment only (Weeks 1-12 for all arms except for Part 2 Deferred Arm which is weeks 16-28).

Part 1:

50 mg grazoprevir + 50 mg elbasvir treatment for 12 weeks, 24 weeks follow-up (Arm 1) 100 mg grazoprevir + 50 mg elbasvir treatment for 12 weeks, 24 weeks follow-up (Arm 2)

Part 2:

Selected dose of grazoprevir + 50 mg elbasvir treatment for 12 weeks, 24 weeks follow-up (Arm 1/Immediate) Placebo treatment for 12 weeks, 4 weeks follow-up, selected dose of grazoprevir + 50 mg elbasvir treatment for 12 weeks, 24 weeks follow-up (Arm 2/Deferred) Selected dose of grazoprevir + 50 mg elbasvir treatment for 12 weeks, 24 weeks follow-up (Arm 3/Cirrhotic)

ELIGIBILITY:
Inclusion Criteria:

* Has documented chronic Japanese HCV genotype (GT) 1 with no evidence of non-typeable or mixed GT infection
* Is treatment-naïve, or intolerant or non-responder to prior anti-HCV interferon (IFN)-based treatment without direct acting antiviral (DAA) therapy, prior IFN-based treatment with DAA therapy, or prior DAA therapy
* Agrees to the use of contraception if a female of reproductive potential

Exclusion Criteria:

* Has evidence of decompensated liver disease manifested by the presence of or history of ascites, esophageal or gastric variceal bleeding, hepatic encephalopathy or other signs or symptoms of advanced liver disease
* Is coinfected with hepatitis B virus or human immunodeficiency virus (HIV)
* Has a history of malignancy ≤5 years prior to signing informed consent except for adequately treated basal cell or squamous cell skin cancer or carcinoma in situ
* Has cirrhosis and liver imaging within 6 months of Day 1 showing evidence of hepatocellular carcinoma (HCC) or is under evaluation for HCC (Part 2 only)
* Has clinically-relevant drug or alcohol abuse within 12 months of screening
* Is a female and is pregnant or breast-feeding, or expecting to conceive or donate eggs from Day 1 and continue throughout treatment and follow-up (or longer if dictated by local regulations)
* Has any of the following conditions:
* Organ transplants (including hematopoietic stem cell transplants) other than cornea and hair
* Poor venous access
* History of gastric surgery (e.g., stapling, bypass) or subject with a history of malabsorption disorders (e.g., celiac sprue disease)
* History of a medical/surgical condition that resulted in hospitalization within the 3 months prior to enrollment, other than for minor elective procedures
* Medical/surgical conditions that may result in a need for hospitalization during the period of the study
* Any medical condition requiring, or likely to require, chronic systemic administration of corticosteroids, TNF antagonists, or other immunosuppressant drugs during the course of the trial
* Has chronic hepatitis not caused by HCV, including but not limited to nonalcoholic steatohepatitis (NASH), drug-induced hepatitis, and autoimmune hepatitis

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 399 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2016-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kumada H, Suzuki Y, Karino Y, Chayama K, Kawada N, Okanoue T, Itoh Y, Mochida S, Toyoda H, Yoshiji H, Takaki S, Yatsuzuka N, Yodoya E, Iwasa T, Fujimoto G, Robertson MN, Black S, Caro L, Wahl J. The combination of elbasvir and grazoprevir for the treatment of chronic HCV infection in Japanese patients: a randomized phase II/III study. J Gastroenterol. 2017 Apr;52(4):520-533. doi: 10.1007/s00535-016-1285-y. Epub 2016 Nov 21. PMID 27873094

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 432 screened, 63 were enrolled and randomized to Part 1 and 336 were enrolled and randomized to Part 2, for a total of 399 randomized.
Groups:
- Part 1 Grazoprevir 50 mg + Elbasvir: Non-cirrhotic participants take 50 mg grazoprevir in combination with 50 mg elbasvir orally (p.o.) once daily (q.d.) for 12 weeks during the blinded period of Part 1 and are followed-up for 24 weeks during the open-label period of Part 1.
- Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir: Non-cirrhotic participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2, and are followed-up for 24 weeks during the open-label period of Part 2.
- Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir: Non-cirrhotic participants take dose-matched placebo p.o. q.d. for 12 weeks during the blinded period of Part 2 followed by a 4-week follow-up. Afterwards, participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks and are followed-up for 24 weeks during the open-label period of Part 2.
- Part 2 Cirrhotic: Grazoprevir + Elbasvir: Cirrhotic participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2, and are followed-up for 24 weeks during the open-label period of Part 2.
Period: Part 1
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Started | 31 | 32 | 0 | 0 | 0
Completed | 31 | 31 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Period: Part 2
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Started | 0 (Participants of Part 1 did not enter Part 2) | 0 (Participants of Part 1 did not enter Part 2) | 227 | 74 | 35
Started Deferred Active Treatment | 0 | 0 | 0 | 73 (1 participant in Deferred Treatment Arm receiving Placebo did not receive Deferred Active Treatment.) | 0
Completed | 0 | 0 | 226 | 71 | 34
Not Completed | 0 | 0 | 1 | 3 | 1
Not completed — Death | 0 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo► Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir | Total
Number analyzed (Participants) | 31 | 32 | 227 | 74 | 35 | 399
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.1 (9.7) | 58.0 (12.5) | 61.1 (12.5) | 60.9 (10.8) | 64.8 (9.2) | 61.1 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 17 | 140 | 53 | 17 | 246
  Male | 12 | 15 | 87 | 21 | 18 | 153

OUTCOME MEASURES:

1. Primary Outcome: Part 2: Percentage of Treatment-naïve Participants in the Immediate Treatment Arm Achieving Sustained Viral Response at 12 Weeks After The End of All Treatment (SVR12)
Description: Blood was drawn from each participant to assess Hepatitis C Virus ribonucleic acid (HCV RNA) plasma levels using the Roche COBAS® Taqman quantitative reverse transcription-polymerase chain reaction (RT-PCR) assay, v2.0, which had a lower limit of quantification (LLoQ) of 1.2 Log IU/mL (15 IU/mL) and a lower limit of detection (LLoD) below 15 IU/ml (no specific value). SVR12 was defined as undetectable HCV RNA (target not detected) at 12 weeks after the end of all study therapy. The Clopper-Pearson method was used to construct 95% confidence intervals (CIs) for the SVR12 rate. The lower limit of the 95% CI was compared to the reference rate of 75%; a lower CI limit that was higher than the reference rate would confirm the primary hypothesis and indicate that that the treatment combination was efficacious. As pre-specified in the protocol, only the Immediate Treatment Arm of Part 2 (treatment naïve participants) was included in the primary efficacy analysis.
Time Frame: 12 weeks after end of all therapy in Part 2 (Study Week 24 of Part 2)
Population: The primary efficacy analysis was assessed in all treatment-naïve participants randomized to the Part 2 Immediate Treatment Arm who received ≥1 dose of study treatment and had any follow-up efficacy measurement. No other arms were analyzed for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir: Non-cirrhotic treatment-naïve participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2, and are followed-up for 24 weeks during the open-label period of Part 2.
- Part 2 Non-cirrhotic Deferred: Placebo: Non-cirrhotic participants take dose-matched placebo p.o. q.d. for 12 weeks during the blinded period of Part 2 followed by a 4-week follow-up.
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Number analyzed (Participants) | 0 | 0 | 149 | 0 | 0
percentage of participants |  |  | 96.6 [92.3 to 98.9] |  |

2. Primary Outcome: Part 1: Percentage of Participants Experiencing an Adverse Event (AE) During Treatment and First 4 Follow-Up Weeks
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, was also an AE. The primary safety evaluation was limited to the initial treatment period through Follow-up Week 4 (FUWK4).
Time Frame: Up to 4 weeks post last dose in Part 1 (Up to total of 16 weeks)
Population: All randomized participants in Part 1 who received ≥1 dose of study treatment and had any safety follow-up data. Data for participants in Part 2 were analyzed and reported separately.
Measure: Number; unit: percentage of participants
Groups:
- Part 1 Grazoprevir 50 mg + Elbasvir: Non-cirrhotic participants take 50 mg grazoprevir in combination with 50 mg elbasvir orally (p.o.) once daily (q.d.) for 12 weeks during the blinded period of Part 1.
- Part 1 Grazoprevir 100 mg + Elbasvir: Non-cirrhotic participants take 100 mg grazoprevir in combination with 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 1.
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir
Number analyzed (Participants) | 31 | 31
percentage of participants | 67.7 | 74.2

3. Primary Outcome: Part 1: Percentage of Participants That Discontinued Treatment Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening (i.e., any clinically significant adverse change in frequency and/or intensity) of a preexisting condition that is temporally associated with the use of the Sponsor's product, was also an AE. The primary safety evaluation was limited to the initial treatment period through FUWK4.
Time Frame: Up to Study Week 12 in Part 1
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir
Number analyzed (Participants) | 31 | 31
percentage of participants | 0.0 | 0.0

4. Secondary Outcome: Part 1: Percentage of Participants Achieving Undetectable HCV RNA Over Time
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® Taqman quantitative RT-PCR assay, v2.0, which had a LLoQ of 1.2 Log IU/mL (15 IU/mL) and a LLoD below 15 IU/ml (no specific value). Undetectable HCV RNA was defined as HCV RNA target not detected. The percentage of participants with undetectable HCV RNA at TW2, TW4, TW12, EOT, FUWK4, FUWK12, and FUWK24 is summarized for each arm. The Clopper-Pearson method was used to construct 95% CIs for SVR rates.
Time Frame: Part 1 Treatment Weeks (TW)2, TW4, TW12, End of Treatment (EOT), FUWK4, FUWK12, FUWK24
Population: All randomized participants in Part 1 who have received ≥1 dose of study treatment and who have any follow-up efficacy measurement. Data for participants in Part 2 were analyzed and reported separately.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir
Number analyzed (Participants) | 31 | 31
percentage of participants
  TW2 | 22.6 [9.6 to 41.1] | 35.5 [19.2 to 54.6]
  TW4 | 77.4 [58.9 to 90.4] | 83.9 [66.3 to 94.5]
  TW12 | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  EOT | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  FUWK4 | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  FUWK12 | 100.0 [88.8 to 100.0] | 96.8 [83.3 to 99.9]
  FUWK24 | 96.8 [83.3 to 99.9] | 96.8 [83.3 to 99.9]

5. Secondary Outcome: Part 1: Percentage of Participants Achieving HCV RNA Below the Lower Limit of Quantitation (<LLoQ) Over Time
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® Taqman quantitative RT-PCR assay, v2.0, which had a LLoQ of 1.2 Log IU/mL (15 IU/mL) and a LLoD below 15 IU/ml (no specific value). Undetectable HCV RNA was defined as HCV RNA target not detected. The percentage of participants with HCV RNA <LLoQ at TW2, TW4, TW12, EOT, FUWK4, FUWK12, and FUWK24 is summarized for each arm. The Clopper-Pearson method was used to construct 95% CIs for SVR rates.
Time Frame: Part 1 TW2, TW4, TW12, EOT, FUWK4, FUWK12, FUWK24
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir
Number analyzed (Participants) | 31 | 31
percentage of participants
  TW2 | 61.3 [42.2 to 78.2] | 71.0 [52.0 to 85.8]
  TW4 | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  TW12 | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  EOT | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  FUWK4 | 100.0 [88.8 to 100.0] | 100.0 [88.8 to 100.0]
  FUWK12 | 100.0 [88.8 to 100.0] | 96.8 [83.3 to 99.9]
  FUWK24 | 100.0 [88.8 to 100.0] | 96.8 [83.3 to 99.9]

6. Primary Outcome: Part 2: Percentage of Participants Experiencing an AE During Initial Treatment and First 4 Follow-Up Weeks
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, was also an AE. The primary safety evaluation was limited to the initial treatment period and first 4 follow-up weeks, and the primary safety statistical analysis compared the percentage of participants with events between the Part 2 Immediate Treatment Arm and the Part 2 Deferred Treatment Arm while receiving placebo.
Time Frame: Up to 4 weeks following initial treatment in Part 2 (Up to total of 16 weeks)
Population: All randomized participants in Part 2 who received ≥1 dose of study treatment and had any safety follow-up data. Participants in the Deferred Arm would have received only placebo treatment up to Study Week 16. Data for participants in Part 1 were analyzed and reported separately.
Measure: Number; unit: percentage of participants
Groups:
- Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir: Non-cirrhotic participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2.
- Part 2 Cirrhotic: Grazoprevir + Elbasvir: Cirrhotic participants take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks during the blinded period of Part 2.
Arm/Group | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Number analyzed (Participants) | 227 | 74 | 35
percentage of participants | 64.8 | 67.6 | 80.0
Statistical Analysis 1: Comparison: Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir vs Part 2 Non-cirrhotic Deferred: Placebo; 95% confidence intervals were provided for between-treatment differences in the percentage of participants with events, comparing participants in the Part 2 Immediate Treatment (Grazoprevir + Elbasvir) Arm with the Part 2 Deferred Treatment (Placebo) Arm during the double blinded period through FUWK4. These analyses were performed using the Miettinen and Nurminen method, an unconditional, asymptotic method; Test type: Superiority or Other; Miettinen and Nurminen Method; Difference in Percentage = -2.8, 95% CI 2-sided [-14.5 to 10.0]

7. Primary Outcome: Part 2: Percentage of Participants That Discontinued Initial Treatment Due to an AE
Description: as for outcome 6
Time Frame: Up to Study Week 12 in Part 2
Population: All randomized participants in Part 2 who received ≥1 dose of study treatment and had any safety follow-up data. Participants in the Deferred Arm would have received only placebo treatment up to Study Week 12. Data for participants in Part 1 were analyzed and reported separately.
Measure: Number; unit: percentage of participants
Groups:
- Part 2 Non-cirrhotic Deferred: Placebo: Non-cirrhotic participants take dose-matched placebo p.o. q.d. for 12 weeks during the blinded period of Part 2.
Arm/Group | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Number analyzed (Participants) | 227 | 74 | 35
percentage of participants | 1.3 | 1.4 | 0.0
Statistical Analysis 1: Comparison: Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir vs Part 2 Non-cirrhotic Deferred: Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; Miettinen and Nurminen Method; Difference in Percentage = -0.0, 95% CI 2-sided [-6.0 to 2.8]

8. Secondary Outcome: Part 2: Percentage of Participants Achieving Undetectable HCV RNA Over Time After Active Treatment
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® Taqman quantitative RT-PCR assay, v2.0, which had a LLoQ of 1.2 Log IU/mL (15 IU/mL) and a LLoD below 15 IU/ml (no specific value). Undetectable HCV RNA was defined as HCV RNA target not detected. The percentage of participants with undetectable HCV RNA at TW2, TW4, TW12, EOT, FUWK4, FUWK12, and FUWK24 is summarized for each arm. Data reported for the Part 2 Deferred Treatment Arm corresponds to the deferred active treatment weeks and subsequent follow-up. The Clopper-Pearson method was used to construct 95% CIs for SVR rates.
Time Frame: Part 2: Active TW2, TW4, TW12, End of Treatment (EOT), FUWK4, FUWK12, FUWK24
Population: All randomized participants in Part 2 who have received ≥1 dose of active study treatment and who have any follow-up efficacy measurement. Data for participants in Part 1 were analyzed and reported separately.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir: During the open-label period of Part 2, non-cirrhotic participants in the Deferred Treatment Arm take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks and are followed-up for 24 weeks.
Arm/Group | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Number analyzed (Participants) | 227 | 73 | 35
percentage of participants
  TW2 | 25.1 [19.6 to 31.3] | 39.7 [28.5 to 51.9] | 11.4 [3.2 to 26.7]
  TW4 | 70.5 [64.1 to 76.3] | 86.3 [76.2 to 93.2] | 65.7 [47.8 to 80.9]
  TW12 | 97.8 [94.9 to 99.3] | 100.0 [95.1 to 100.0] | 100.0 [90.0 to 100.0]
  EOT | 98.7 [96.2 to 99.7] | 100.0 [95.1 to 100.0] | 100.0 [90.0 to 100.0]
  FUWK4 | 98.2 [95.5 to 99.5] | 100.0 [95.1 to 100.0] | 97.1 [85.1 to 99.9]
  FUWK12 | 96.5 [93.2 to 98.5] | 95.9 [88.5 to 99.1] | 97.1 [85.1 to 99.9]
  FUWK24 | 96.5 [93.2 to 98.5] | 95.9 [88.5 to 99.1] | 94.3 [80.8 to 99.3]

9. Secondary Outcome: Part 2: Percentage of Participants Achieving HCV RNA <LLoQ Over Time After Active Treatment
Description: Blood was drawn from each participant to assess HCV RNA plasma levels using the Roche COBAS® Taqman quantitative RT-PCR assay, v2.0, which had a LLoQ of 1.2 Log IU/mL (15 IU/mL) and a LLoD below 15 IU/ml (no specific value). Undetectable HCV RNA was defined as HCV RNA target not detected. The percentage of participants with HCV RNA <LLoQ at TW2, TW4, TW12, EOT, FUWK4, FUWK12, and FUWK24 is summarized for each arm. Data reported for the Part 2 Deferred Treatment Arm corresponds to the deferred active treatment weeks and subsequent follow-up. The Clopper-Pearson method was used to construct 95% CIs for SVR rates.
Time Frame: Part 2: Active TW2, TW4, TW12, End of Treatment (EOT), FUWK4, FUWK12, FUWK24
Population: as for outcome 8
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Number analyzed (Participants) | 227 | 73 | 35
percentage of participants
  TW2 | 60.8 [54.1 to 67.2] | 69.9 [58.0 to 80.1] | 60.0 [42.1 to 76.1]
  TW4 | 96.0 [92.6 to 98.2] | 98.6 [92.6 to 100.0] | 94.3 [80.8 to 99.3]
  TW12 | 98.7 [96.2 to 99.7] | 100.0 [95.1 to 100.0] | 100.0 [90.0 to 100.0]
  EOT | 99.6 [97.6 to 100.0] | 100.0 [95.1 to 100.0] | 100.0 [90.0 to 100.0]
  FUWK4 | 98.2 [95.5 to 99.5] | 100.0 [95.1 to 100.0] | 97.1 [85.1 to 99.9]
  FUWK12 | 96.5 [93.2 to 98.5] | 97.3 [90.5 to 99.7] | 97.1 [85.1 to 99.9]
  FUWK24 | 96.5 [93.2 to 98.5] | 95.9 [88.5 to 99.1] | 97.1 [85.1 to 99.9]

ADVERSE EVENTS:
Time Frame: Part 1: Up to a total of 36 weeks Part 2: Up to a total of 52 weeks
Description: All randomized participants who received ≥1 dose of study treatment and had any safety follow-up data. AEs were reported by the treatment that participants were receiving at the time of the event; AEs for Deferred Arm reported separately for placebo and active treatment. Part 1 database=MedDRA 18.1, Part 2 database=MedDRA 19.0
Groups:
- Part 2 Non-cirrhotic Deferred: Placebo: Non-cirrhotic participants in the Deferred Treatment Arm take dose-matched placebo p.o. q.d. for 12 weeks during the blinded period of Part 2 followed by a 4-week follow-up.
- Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir: During the open-label period, non-cirrhotic participants in the Deferred Treatment Arm take 100 mg grazoprevir and 50 mg elbasvir p.o. q.d. for 12 weeks and are followed-up for 24 weeks. One participant who received placebo during the blinded period did not receive active treatment during the open-label period.
Arm/Group | Part 1 Grazoprevir 50 mg + Elbasvir | Part 1 Grazoprevir 100 mg + Elbasvir | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir | Part 2 Non-cirrhotic Deferred: Placebo | Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir | Part 2 Cirrhotic: Grazoprevir + Elbasvir
Serious Adverse Events (participants affected / at risk) | 2/31 | 1/31 | 19/227 | 1/74 | 2/73 | 3/35
Other Adverse Events (participants affected / at risk) | 16/31 | 17/31 | 109/227 | 27/74 | 42/73 | 27/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Grazoprevir 50 mg + Elbasvir (N=31) | Part 1 Grazoprevir 100 mg + Elbasvir (N=31) | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir (N=227) | Part 2 Non-cirrhotic Deferred: Placebo (N=74) | Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir (N=73) | Part 2 Cirrhotic: Grazoprevir + Elbasvir (N=35)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac sarcoidosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign anorectal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lead dislodgement (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — appears under "Product Issues" in MedDRA v. 19.0
Ureterolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 Grazoprevir 50 mg + Elbasvir (N=31) | Part 1 Grazoprevir 100 mg + Elbasvir (N=31) | Part 2 Non-cirrhotic Immediate: Grazoprevir + Elbasvir (N=227) | Part 2 Non-cirrhotic Deferred: Placebo (N=74) | Part 2 Non-cirrhotic Deferred: Grazoprevir + Elbasvir (N=73) | Part 2 Cirrhotic: Grazoprevir + Elbasvir (N=35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Conjunctival haemorrhage (Eye disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 6 (6) | 1 (1) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 11 (11) | 3 (3) | 4 (4) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (2) | 12 (14) | 2 (3) | 6 (6) | 3 (3)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0) | 7 (7) | 3 (5) | 5 (6) | 2 (2)
Pyrexia (General disorders) | 3 (3) | 1 (2) | 3 (3) | 1 (1) | 3 (3) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 8 (9) | 1 (1) | 6 (6) | 1 (1)
Nasopharyngitis (Infections and infestations) | 8 (12) | 11 (12) | 47 (56) | 12 (18) | 20 (25) | 8 (11)
Periodontitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
Accidental overdose (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 5 (5) | 1 (1) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 12 (12) | 1 (1) | 3 (3) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 10 (10) | 2 (3) | 3 (3) | 6 (6)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0) | 7 (7) | 4 (4) | 3 (4) | 1 (1)
Protein urine present (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 8 (8) | 0 (0) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 5 (6) | 3 (3) | 11 (13) | 2 (2) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 9 (10) | 1 (1) | 0 (0) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator or sub-investigators may publicly present the academic accomplishment acquired from the Study at a specialized academic meeting or research conference. The Sponsor may freely use the information acquired from the Study for the purpose of marketing authorization application of the test drug.